CLINICAL TRIAL: NCT00199290
Title: A Phase 2, Randomized, Double Blind, Placebo-Controlled, Parallel Group Study to Evaluate the Efficacy and the Safety of Trafermin in Patients With Marginal Periodontitis in Japan
Brief Title: A Phase2 Clinical Trial of Trafermin in Patients With Marginal Periodontitis in Japan
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kaken Pharmaceutical (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KCB-1D-02
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2008-02-05 (Estimated); Status verified 2008-02

CONDITIONS: Periodontitis
Keywords: Trafermin; Periodontitis
MeSH Terms: conditions — Periodontitis | interventions — trafermin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- P (Placebo Comparator)
  Interventions: Drug: Trafermin (genetical recombination)
- L (Experimental): low dose (0.2 %)
  Interventions: Drug: Trafermin (genetical recombination)
- M (Experimental): medium dose (0.3 %)
  Interventions: Drug: Trafermin (genetical recombination)
- H (Experimental): high dose (0.4 %)
  Interventions: Drug: Trafermin (genetical recombination)

INTERVENTIONS:
Drug: Trafermin (genetical recombination)

SUMMARY:
This study is designed to evaluate the efficacy and the safety of Trafermin(recombinant human basic fibroblast growth factor: rhbFGF) in Japanese patients with marginal periodontitis, in order to verify the superiority of Trafermin to placebo, and to determine the recommended therapeutic dose.

ELIGIBILITY:
Inclusion Criteria:

The patient with marginal periodontitis intend to conduct a flap operation(modified Widman) must meet the following criteria:

* Alveolar bone defect diagnosed by radiography.
* Mobility of teeth must be <=2 and the width of attached gingiva is suitable for GTR(guided tissue regeneration) method.
* Males and females, >=20 years of age.

Exclusion Criteria:

Patients will be excluded from the study if any of the following conditions are present:

* Concomitant administration of adrenal cortical steroid within 4weeks of treatment in the trial.
* Current or previous history of gingival overgrowth by drugs.
* Current or previous history of cancer or malignant tumour.
* Presence of diabetes mellitus(HbA1c>=6.5%)
* Presence of malnutrition(serum albumin<=2g/dL)
* Pregnancy or lactation

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 267 (Actual)
Dates: Start 2005-08; Primary Completion 2007-07 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
rate of increase in alveolar bone height | 36 weeks after administration

SECONDARY OUTCOMES:
clinical attachment level regained | 36 weeks after administration
time course of increase rate in alveolar bone height | within 36 weeks after administration
time course of clinical attachment level regained | within 36 weeks after administration
occurrence and level of adverse reaction | within 36 weeks after administration
serum anti-Trafermin antibody level | within 4 weeks
serum Trafermin level | within 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Makoto Tamura, Ph.D, Study Director — Kaken Pharmaceutical Co., Ltd.
Locations (22):
- Japan (22):
  - Kaken Investigational Site, Nagoya, Aichi-ken
  - Kaken Investigational Site, Chiba, Chiba
  - Kaken Investigational Site, Matsudo, Chiba
  - Kaken Investigational Site, Fukuoka, Fukuoka
  - Kaken Investigational Site, Kitakyushu, Fukuoka
  - Kaken Investigational Site, Mizuho, Gifu
  - Kaken Investigational Site, Hiroshima, Hiroshima
  - Kaken Investigational Site, Ishikari-gun, Hokkaido
  - Kaken Investigational Site, Sapporo, Hokkaido
  - Kaken Investigational Site, Morioka, Iwate
  - Kaken Investigational Site, Kagoshima, Kagoshima-ken
  - Kaken Investigational Site, Yokohama, Kanagawa
  - Kaken Investigational Site, Sendai, Miyagi
  - Kaken Investigational Site, Nagasaki, Nagasaki
  - Kaken Investigational Site, Niigata, Niigata
  - Kaken Investigational Site, Okayama, Okayama-ken
  - Kaken Investigational Site, Suita, Osaka
  - Kaken Investigational Site, Tokushima, Tokushima
  - Kaken Investigational Site, Bunkyo-ku, Tokyo
  - Kaken Investigational Site, Chiyoda-ku, Tokyo
  - Kaken Investigational Site, Machida, Tokyo
  - Kaken Investigational Site, Sinjyuku-ku, Tokyo